CLINICAL TRIAL: NCT02877745
Title: ImpaCt of Sleep-disOrdered breathiNg on Atrial Fibrillation and Perioperative complicationS In Patients unDERgoing Coronary Artery Bypass graFting Surgery
Brief Title: Sleep-disordered Breathing and Perioperative Atrial Fibrillation in Cardiac Surgery
Acronym: CONSIDER-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Michael Arzt (Other)
Responsible Party: Sponsor-Investigator, Michael Arzt, Coordinating Investigator, University Hospital Regensburg
Organization: University Hospital Regensburg (Other)
Other Study IDs: 3643420
Record Dates: First submitted 2016-07-31; First posted 2016-08-24 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Elective Coronary Artery Bypass Grafting (CABG) Surgery; Coronary Artery Disease; Sleep-disordered Breathing (SDB); Atrial Fibrillation
MeSH Terms: conditions — Coronary Artery Disease; Sleep Apnea Syndromes; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- no SDB: apnea-hyponea index <15/hour
  Interventions: Other: Stratification, no intervention
- SDB: apnea-hyponea index >=15/hour
  Interventions: Other: Stratification, no intervention

INTERVENTIONS:
Other: Stratification, no intervention

SUMMARY:
In patients undergoing elective coronary artery bypass grafting (CABG) surgery, coronary artery disease, sleep-disordered breathing (SDB), atrial fibrillation (AF) perioperative atrial fibrillation and complications will be assessed. The primary objective is to determine, whether SDB patients have a higher rate of Major Adverse Cardiac and Cerebrovascular Events (MACCE) within 30 days after surgery compared to those without SDB.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective CABG surgery at the Department of Cardiac and Thoracic Surgery, University Hospital Regensburg.
* Written informed consent

Exclusion Criteria:

* Preoperative use of inotropes or intra aortic balloon pump
* Severe obstructive pulmonary disease
* Patients on oxygen therapy, nocturnal positive airway pressure support or mechanical ventilation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be consecutive patients undergoing elective CABG surgery in stable hemodynamic condition. Only individuals who can give written informed consent will be included. Gender distribution will be according to the gender distribution of patients undergoing elective CABG surgery, since consecutive patients without gender selection will be studied.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2016-07; Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 30 days
  periprocedural and late myocardial infarction (MI), non-fatal stroke and transitory ischemic attack (TIA) as well as all-cause mortality

SECONDARY OUTCOMES:
postoperative atrial fibrillation (POAF) | 30 days after CABG surgery
  assessed by ECG
Stroke | within 1 year after CABG surgery
  assessed by questionnaire
MACCE | within 1 and 2 years after CABG surgery
  assessed by questionnaire
Major pulmonary complications | within 30 days as well as 1 and 2 years
  assessed by questionnaire

OTHER OUTCOMES:
peri- and postoperative respiratory complications (difficult intubation, hypoxemia, respiratory failure, use of extracorporal mechanical oxygenation device) | 30 days after CABG surgery
  Assessed from standardized routine clinical records
peri- and postoperative hemodynamic instability and heart failure | 30 days after CABG surgery
  (medical records)
postoperative enzymatic myocardial injury | 30 days after CABG surgery
  (medical records)
postoperative acute kidney injury | 30 days after CABG surgery
  (medical records)
postoperative delirium | 30 days after CABG surgery
  (Questionnaire)
general quality of life | 30 days after CABG surgery
  (EuroQol - Questionnaire)
disease specific quality of life | 30 days after CABG surgery
  (Atrial Fibrillation Effect on Quality of Life - Questionnaire)
disease specific quality of life | 30 days after CABG surgery
  (Seattle Angina Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Lars S Maier, MD, Principal Investigator — University Hospital Regensburg
Locations (1):
- Department of Internal Medicine II, University Hospital, Regensburg, Germany

REFERENCES:
- [Derived] Tafelmeier M, Blagoeva VG, Trum M, Hegner P, Floerchinger B, Camboni D, Creutzenberg M, Zeman F, Schmid C, Maier LS, Wagner S, Linz D, Baumert M, Arzt M. Predictors of Nocturnal Hypoxemic Burden in Patients Undergoing Elective Coronary Artery Bypass Grafting Surgery. Biomedicines. 2023 Sep 28;11(10):2665. doi: 10.3390/biomedicines11102665. PMID 37893039
- [Derived] Hegner P, Lebek S, Tafelmeier M, Camboni D, Schopka S, Schmid C, Maier LS, Arzt M, Wagner S. Sleep-disordered breathing is independently associated with reduced atrial connexin 43 expression. Heart Rhythm. 2021 Dec;18(12):2187-2194. doi: 10.1016/j.hrthm.2021.09.009. Epub 2021 Sep 10. PMID 34517118
- [Derived] Lebek S, Hegner P, Tafelmeier M, Rupprecht L, Schmid C, Maier LS, Arzt M, Wagner S. Female Patients With Sleep-Disordered Breathing Display More Frequently Heart Failure With Preserved Ejection Fraction. Front Med (Lausanne). 2021 May 28;8:675987. doi: 10.3389/fmed.2021.675987. eCollection 2021. PMID 34124106
- [Derived] Tafelmeier M, Luft L, Zistler E, Floerchinger B, Camboni D, Creutzenberg M, Zeman F, Schmid C, Maier LS, Wagner S, Arzt M. Central Sleep Apnea Predicts Pulmonary Complications After Cardiac Surgery. Chest. 2021 Feb;159(2):798-809. doi: 10.1016/j.chest.2020.07.080. Epub 2020 Aug 13. PMID 32798522
- [Derived] Lebek S, Pichler K, Reuthner K, Trum M, Tafelmeier M, Mustroph J, Camboni D, Rupprecht L, Schmid C, Maier LS, Arzt M, Wagner S. Enhanced CaMKII-Dependent Late INa Induces Atrial Proarrhythmic Activity in Patients With Sleep-Disordered Breathing. Circ Res. 2020 Feb 28;126(5):603-615. doi: 10.1161/CIRCRESAHA.119.315755. Epub 2020 Jan 6. PMID 31902278
- [Derived] Tafelmeier M, Knapp M, Lebek S, Floerchinger B, Camboni D, Creutzenberg M, Wittmann S, Zeman F, Schmid C, Maier LS, Wagner S, Arzt M. Predictors of delirium after cardiac surgery in patients with sleep disordered breathing. Eur Respir J. 2019 Aug 8;54(2):1900354. doi: 10.1183/13993003.00354-2019. Print 2019 Aug. PMID 31109986